CLINICAL TRIAL: NCT02198430
Title: Multidisciplinary Assessment of the Physical, Functional and Psychosocial Alterations in Patients With Hemophilia. An Observational Study.
Brief Title: Multidisciplinary Evaluation of Patients With Hemophilia
Acronym: HOLISTIC
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, ANA TORRES-ORTUÑO, PhD, Universidad de Murcia
Other Study IDs: Hemo-HOLISTIC; HOLISTIC
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-06

CONDITIONS: Haemophilia
Keywords: Haemophilia; Arthropathy; Range of motion; Strength; Proprioception; Gait; Quality of Life.
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with haemophilia recruited for multidisciplinary assessment of the main physical, functional and psychosocial variables.
- Control group: Children without hemophilia

SUMMARY:
Multidisciplinary assessment of the physical, functional and psychosocial alterations in patients with hemophilia around the country. The aims of this study are:

* Descriptive study of joint involvement in hemophilia patients with and without a history of hemarthrosis.
* Descriptive study of the alterations of periarticular muscle strength as a result of acute processes or the development of chronic articular sequelae.
* Descriptive study of biomechanical changes in lower limb joints and their impact on gait in patients with hemophilia.
* Descriptive study of the joint space, regarding hemarthrosis and synovitis, intraarticular by ultrasonography.
* Descriptive study of the relationship between skeletal muscle pathology in patients with hemophilia and their perceptions of it and their quality of life.

DETAILED DESCRIPTION:
Observational study that will allow us:

Analyze and evaluate the skeletal muscle of patients with hemophilia involvement.

Describe the periarticular muscular deficit, depending on the degree of injury, age, presence of inhibitors and the development of physical activity.

Identify the relationship between the functional deficit by clinical assessment performed with the use of validated scales measure force production with patients.

Observe the presence of joint bleeds in children with hemophilia and synovial hypertrophy developing therein.

Detect biomechanical abnormalities of the lower limbs and their impact on gait in patients with hemophilia.

Assess the factors that influence the perception of illness and quality of life of patients with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A and B.
* Patients of all ages (pediatric, adolescents, youth and adults).
* With or without joint involvement clinically diagnosed, and with or without a previous history of hemarthrosis joint loading.
* Patients with or without inhibitors.

Exclusion Criteria:

* Patients without prior walking capacity.
* Patients diagnosed with other congenital coagulopathy (von Willebrand disease, etc..).
* Patients with neurological or cognitive impairments that prevent understanding the questionnaires and physical tests.

Ages: 8 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with haemophilia attending hemophilia shelters organized by the Federación Española de Hemofilia (Fedhemo) in the Centro de Formación Permanente en Hemofilia La Charca (Murcia, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Catholic University San Antonio of Murcia
Locations (1):
- Universidad de Murcia, Murcia, Murcia, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients | Control Group
Started | 53 | 51
Completed | 53 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Control Group | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.08 (1.36) | 9.78 (1.22) | 10.04 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 51 | 104
Region of Enrollment [Number; unit: participants]
  Spain | 53 | 51 | 104

OUTCOME MEASURES:

1. Primary Outcome: Assess the Joint Damage
Description: Measurement with Haemophilia Joint Health Score 2.1 (HJHS)
Time Frame: Screening visit
Population: Haemophilia Joint Health Score assesses joint health in patients with hemophilia. It consists of eight dimensions: swelling, muscular atrophy, crepitation and range of motion, joint pain, strength, motion and axial alignment. The score range is from 0 to 24 points (a score of 0 indicates no joint damage. The higher the score, the higher).
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Patients | Control Group
Number analyzed (Participants) | 53 | 51
points | 0.36 (0.84) | 0 (0)

2. Primary Outcome: Assess the Perception of Quality of Life
Description: Measurement through the Child health profile (Childhood Health and Illness Perception; CHIP-CE).
Time Frame: Screening visit
Population: The score ranges from 0 (poor QoL) to 100 points (good perception of QoL).
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Patients | Control Group
Number analyzed (Participants) | 53 | 51
points | 38.32 (4.72) | 37.55 (5.91)

3. Secondary Outcome: Assessment of Clinical Patient Variables
Description: Hemophilia type measuring (A or B)
Time Frame: Screening visit
Measure: Number; unit: Percentage of Participants with Hemophil
Arm/Group | Patients | Control Group
Number analyzed (Participants) | 53 | 51
Percentage of Participants with Hemophil | 92.5 | 0

4. Secondary Outcome: Measure of Weight
Description: Measure of weight
Time Frame: Screening visit (pretreatment assessment)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Patients | Control Group
Number analyzed (Participants) | 53 | 51
Kg | 41.59 (11.82) | 39.36 (9.64)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Patients | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less